CLINICAL TRIAL: NCT02924129
Title: A Prospective, Multicenter, Randomized Double-blind Study Examining the Safety and Efficacy of Using the Evoke™ Spinal Cord Stimulator (SCS) System With Feedback to Treat Patients With Chronic Pain of the Trunk and/or Limbs.
Brief Title: Safety and Efficacy Study of the Evoke™ SCS System With Feedback vs. Conventional Stimulation
Acronym: EVOKE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saluda Medical Americas, Inc. (Industry)
Responsible Party: Sponsor
Organization: Saluda Medical Pty Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCLSH1503
Record Dates: First submitted 2016-09-30; First posted 2016-10-05 (Estimated); Results first posted 2021-05-25 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Chronic Pain; Back Pain; Pain
Keywords: Chronic Pain; Back Pain; Leg Pain; Pain; Neurologic Manifestations; Nervous System Diseases; Signs and Symptoms; SCS; Closed Loop
MeSH Terms: conditions — Chronic Pain; Back Pain; Pain; Neurologic Manifestations; Nervous System Diseases; Signs and Symptoms | interventions — Spinal Cord Stimulation; Drug Delivery Systems

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Evoke SCS with Feedback (Experimental): closed-loop/automatic stimulation
  Interventions: Device: Evoke Spinal Cord Stimulator (SCS) System
- Evoke SCS with Conventional (Active Comparator): open-loop/manual stimulation
  Interventions: Device: Evoke Spinal Cord Stimulator (SCS) System

INTERVENTIONS:
Device: Evoke Spinal Cord Stimulator (SCS) System — Spinal Cord Stimulation that measures and records evoked compound action potentials (ECAPs).

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the Saluda Medical Evoke SCS System with feedback control to treat chronic pain of the trunk and/or limbs.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female between the ages of 18 and 80 years.
* Have been diagnosed with chronic, intractable pain of the trunk and/or limbs, which has been refractory to conservative therapy for a minimum of 6 months.
* Be an appropriate candidate for an SCS trial and the surgical procedures required in this study based on the clinical judgment of the Investigator.
* Be willing and capable of giving informed consent and able to comply with study-related requirements, procedures, and visits.

Exclusion Criteria:

* Have a medical condition or pain in other area(s), not intended to be treated with SCS, that could interfere with study procedures, accurate pain reporting, and/or confound evaluation of study endpoints, as determined by the Investigator.
* Have evidence of an active disruptive psychological or psychiatric disorder or other known condition significant enough to impact perception of pain, compliance of intervention, and/or ability to evaluate treatment outcomes.
* Have an existing drug pump and/or SCS system or another active implantable device such as a pacemaker, deep brain stimulator (DBS), or sacral nerve stimulator (SNS).
* Have prior experience with SCS.
* Have an active systemic infection or local infection in the area of the surgical site.
* Be pregnant or nursing (if female and sexually active, subject must be using a reliable form of birth control, be surgically sterile, or be at least 2 years post-menopausal).
* Be concomitantly participating in another clinical study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2017-01-27 (Actual); Primary Completion 2018-06-21 (Actual); Study Completion 2022-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dan Brounstein, MBA, Study Director — Saluda Medical Americas, Inc.
Locations (16):
- United States (16):
  - Hope Research Institute, Phoenix, Arizona
  - Arizona Pain Specialists, Scottsdale, Arizona
  - Summit Pain Alliance, Santa Rosa, California
  - Thrive Clinic, Santa Rosa, California
  - IPM Medical Group, Walnut Creek, California
  - Pain Management Associates, Lee's Summit, Missouri
  - Premier Pain Centers, Shrewsbury, New Jersey
  - Ainsworth Institute of Pain Management, New York, New York
  - Center for Clinical Research, Winston-Salem, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Integrated Pain Solutions, Columbus, Ohio
  - St. Luke's University Health Network, Bethlehem, Pennsylvania
  - Delaware Valley Pain & Spine Institute, Feasterville-Trevose, Pennsylvania
  - Center for Pain Relief, Charleston, West Virginia
  - Advanced Pain Management, Greenfield, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mekhail NA, Levy RM, Deer TR, Kapural L, Li S, Amirdelfan K, Pope JE, Hunter CW, Rosen SM, Costandi SJ, Falowski SM, Burgher AH, Gilmore CA, Qureshi FA, Staats PS, Scowcroft J, McJunkin T, Carlson J, Kim CK, Yang MI, Stauss T, Petersen EA, Hagedorn JM, Rauck R, Kallewaard JW, Baranidharan G, Taylor RS, Poree L, Brounstein D, Duarte RV, Gmel GE, Gorman R, Gould I, Hanson E, Karantonis DM, Khurram A, Leitner A, Mugan D, Obradovic M, Ouyang Z, Parker J, Single P, Soliday N; EVOKE Study Group. ECAP-controlled closed-loop versus open-loop SCS for the treatment of chronic pain: 36-month results of the EVOKE blinded randomized clinical trial. Reg Anesth Pain Med. 2024 May 7;49(5):346-354. doi: 10.1136/rapm-2023-104751. PMID 37640452
- [Derived] Kapural L, Mekhail NA, Costandi S, Gilmore C, Pope JE, Li S, Hunter CW, Poree L, Staats PS, Taylor RS, Eldabe S, Kallewaard JW, Thomson S, Petersen EA, Sayed D, Deer TR, Antony A, Budwany R, Leitner A, Soliday N, Duarte RV, Levy RM. Durable multimodal and holistic response for physiologic closed-loop spinal cord stimulation supported by objective evidence from the EVOKE double-blind randomized controlled trial. Reg Anesth Pain Med. 2024 Apr 2;49(4):233-240. doi: 10.1136/rapm-2023-104639. PMID 37491149
- [Derived] Costandi S, Kapural L, Mekhail NA, Jotwani R, Bertisch SM, Li S, Petersen E, Abejon D, Poree L, Ouyang Z, Venkatesan L, Mekhail MN, Gilligan CJ. Impact of Long-Term Evoked Compound Action Potential Controlled Closed-Loop Spinal Cord Stimulation on Sleep Quality in Patients With Chronic Pain: An EVOKE Randomized Controlled Trial Study Subanalysis. Neuromodulation. 2023 Jul;26(5):1030-1038. doi: 10.1016/j.neurom.2022.10.050. Epub 2022 Nov 25. PMID 36437161
- [Derived] Falowski SM, Kim CH, Obradovic M, Parker JL. A Prospective Multicenter Case Series Utilizing Intraoperative Neuromonitoring With Evoked Compound Action Potentials to Confirm Spinal Cord Stimulation Lead Placement. Neuromodulation. 2022 Jul;25(5):724-730. doi: 10.1016/j.neurom.2021.11.014. Epub 2022 Jan 26. PMID 35088735
- [Derived] Mekhail N, Levy RM, Deer TR, Kapural L, Li S, Amirdelfan K, Hunter CW, Rosen SM, Costandi SJ, Falowski SM, Burgher AH, Pope JE, Gilmore CA, Qureshi FA, Staats PS, Scowcroft J, Carlson J, Kim CK, Yang MI, Stauss T, Poree L; Evoke Study Group. Long-term safety and efficacy of closed-loop spinal cord stimulation to treat chronic back and leg pain (Evoke): a double-blind, randomised, controlled trial. Lancet Neurol. 2020 Feb;19(2):123-134. doi: 10.1016/S1474-4422(19)30414-4. Epub 2019 Dec 20. PMID 31870766

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Evoke SCS With Feedback | Evoke SCS With Conventional
Started | 67 | 67
Completed | 62 | 63
Not Completed | 5 | 4
Not completed — Adverse Event Unrelated to Device or Stimulation | 2 | 1
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Missed Visit | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Evoke SCS With Feedback | Evoke SCS With Conventional | Total
Number analyzed (Participants) | 67 | 67 | 134
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (9.7) | 55.9 (11.6) | 55.2 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 32 | 65
  Male | 34 | 35 | 69
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 6 | 9
  Not Hispanic or Latino | 64 | 61 | 125
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 6 | 8
  White | 63 | 59 | 122
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 67 | 67 | 134

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Composite Endpoint Success
Description: The primary endpoint is a composite endpoint. A success is defined as a reduction in overall trunk and limb VAS pain score greater than or equal to 50 percent and no increase in baseline pain medication. VAS = Visual Analog Scale, from 0 to 100 mm, where 0 = no pain and 100 = worst imaginable pain.
Time Frame: 3 months
Population: Intention-to-Treat (ITT), which included randomized patients with either known endpoint status or classified as a presumed non-responder (i.e., <50% reduction in overall pain at trial or withdrew due to a device- or stimulation-related adverse event), and therefore imputed as a failure.
Measure: Count of Participants; unit: Participants
Arm/Group | Evoke SCS With Feedback | Evoke SCS With Conventional
Number analyzed (Participants) | 62 | 63
Participants | 51 | 38
Statistical Analysis 1: Comparison: Evoke SCS With Feedback vs Evoke SCS With Conventional; Test type: Non-Inferiority — non-inferiority margin (δ) of 10%; p < 0.001, normal approximation to the binomial — Significance threshold (α) of 0.05

2. Secondary Outcome: Percent Change From Baseline in Leg Pain VAS Score
Description: VAS = Visual Analog Scale, from 0 to 100 mm, where 0 = no pain and 100 = worst imaginable pain.
Time Frame: 3 months
Population: Intention-to-Treat (ITT)
Measure: Mean (Standard Deviation); unit: percentage change in VAS leg pain
Arm/Group | Evoke SCS With Feedback | Evoke SCS With Conventional
Number analyzed (Participants) | 62 | 63
percentage change in VAS leg pain | 76.8 (28.3) | 67.8 (35.5)
Statistical Analysis 1: Comparison: Evoke SCS With Feedback vs Evoke SCS With Conventional; Test type: Non-Inferiority — non-inferiority margin (δ) of 10%; p < 0.001, t-test, 2 sided — significance threshold (α) of 0.05; Mean Difference (Final Values) = 9.0, 95% CI 2-sided [-2.4 to 20.4]

3. Secondary Outcome: Percent Change From Baseline in Back Pain VAS Score
Description: VAS = Visual Analog Scale, from 0 to 100 mm, where 0 = no pain and 100 = worst imaginable pain.
Time Frame: 3 months
Population: Intention-to-Treat (ITT)
Measure: Mean (Standard Deviation); unit: percentage change in VAS back pain
Arm/Group | Evoke SCS With Feedback | Evoke SCS With Conventional
Number analyzed (Participants) | 62 | 63
percentage change in VAS back pain | 72.1 (29.4) | 57.5 (36.4)
Statistical Analysis 1: Comparison: Evoke SCS With Feedback vs Evoke SCS With Conventional; Test type: Non-Inferiority — non-inferiority margin (δ) of 10%; p < 0.001, t-test, 2 sided — significance threshold (α) of 0.05; Mean Difference (Final Values) = 14.6, 95% CI 2-sided [2.9 to 26.3]

4. Secondary Outcome: Proportion of Subjects With Greater Than or Equal to 80% Reduction From Baseline in Overall Trunk and Limb Pain VAS Score
Description: VAS = Visual Analog Scale, from 0 to 100 mm, where 0 = no pain and 100 = worst imaginable pain.
Time Frame: 3 months
Population: Intention-to-Treat (ITT)
Measure: Count of Participants; unit: Participants
Arm/Group | Evoke SCS With Feedback | Evoke SCS With Conventional
Number analyzed (Participants) | 62 | 63
Participants | 36 | 27
Statistical Analysis 1: Comparison: Evoke SCS With Feedback vs Evoke SCS With Conventional; Test type: Non-Inferiority — non-inferiority margin (δ) of 10%; p = 0.002, normal approximation to the binomial — significance threshold (α) of 0.05

5. Secondary Outcome: Proportion of Subjects With Greater Than or Equal to 50% Reduction From Baseline in Back Pain VAS Score
Description: VAS = Visual Analog Scale, from 0 to 100 mm, where 0 = no pain and 100 = worst imaginable pain
Time Frame: 3 months
Population: Intention-to-Treat (ITT)
Measure: Count of Participants; unit: Participants
Arm/Group | Evoke SCS With Feedback | Evoke SCS With Conventional
Number analyzed (Participants) | 62 | 63
Participants | 50 | 36
Statistical Analysis 1: Comparison: Evoke SCS With Feedback vs Evoke SCS With Conventional; Test type: Non-Inferiority — non-inferiority margin (δ) of 10%; p < 0.001, normal approximation to the binomial — significance threshold (α) of 0.05

6. Secondary Outcome: Number of Participants With Composite Endpoint Success
Description: as for outcome 1
Time Frame: 12 months
Population: Intention-to-Treat (ITT)
Measure: Count of Participants; unit: Participants
Arm/Group | Evoke SCS With Feedback | Evoke SCS With Conventional
Number analyzed (Participants) | 59 | 59
Participants | 49 | 36
Statistical Analysis 1: Comparison: Evoke SCS With Feedback vs Evoke SCS With Conventional; Test type: Non-Inferiority — non-inferiority margin (δ) of 10%; p < 0.001, normal approximation to the binomial — significance threshold (α) of 0.05

7. Secondary Outcome: Percent Change From Baseline in Leg Pain VAS Score
Description: VAS = Visual Analog Scale, from 0 to 100 mm, where 0 = no pain and 100 = worst imaginable pain
Time Frame: 12 months
Population: Intention-to-Treat (ITT)
Measure: Mean (Standard Deviation); unit: percentage change in VAS leg pain
Arm/Group | Evoke SCS With Feedback | Evoke SCS With Conventional
Number analyzed (Participants) | 59 | 59
percentage change in VAS leg pain | 72.9 (31.0) | 62.1 (37.5)
Statistical Analysis 1: Comparison: Evoke SCS With Feedback vs Evoke SCS With Conventional; Test type: Non-Inferiority — non-inferiority margin (δ) of 10%; p < 0.001, t-test, 2 sided — significance threshold (α) of 0.05; Mean Difference (Final Values) = 10.7, 95% CI 2-sided [-1.8 to 23.3]

8. Secondary Outcome: Percent Change From Baseline in Back Pain VAS Score
Description: VAS = Visual Analog Scale, from 0 to 100 mm, where 0 = no pain and 100 = worst imaginable pain
Time Frame: 12 months
Population: Intention-to-Treat (ITT)
Measure: Mean (Standard Deviation); unit: percentage change in VAS back pain
Arm/Group | Evoke SCS With Feedback | Evoke SCS With Conventional
Number analyzed (Participants) | 59 | 59
percentage change in VAS back pain | 69.4 (30.6) | 54.0 (39.5)
Statistical Analysis 1: Comparison: Evoke SCS With Feedback vs Evoke SCS With Conventional; Test type: Non-Inferiority — non-inferiority margin (δ) of 10%; p < 0.001, t-test, 2 sided — significance threshold (α) of 0.05; Mean Difference (Final Values) = 15.4, 95% CI 2-sided [2.5 to 28.3]

9. Secondary Outcome: Proportion of Subjects With Greater Than or Equal to 80% Reduction From Baseline in Overall Trunk and Limb Pain VAS Score
Description: VAS = Visual Analog Scale, from 0 to 100 mm, where 0 = no pain and 100 = worst imaginable pain
Time Frame: 12 months
Population: Intention-to-Treat (ITT)
Measure: Count of Participants; unit: Participants
Arm/Group | Evoke SCS With Feedback | Evoke SCS With Conventional
Number analyzed (Participants) | 59 | 59
Participants | 33 | 22
Statistical Analysis 1: Comparison: Evoke SCS With Feedback vs Evoke SCS With Conventional; Test type: Non-Inferiority — non-inferiority margin (δ) of 10%; p < 0.001, normal approximation to the binomial

10. Secondary Outcome: Proportion of Subjects With Greater Than or Equal to 50% Reduction From Baseline in Back Pain VAS Score
Description: VAS = Visual Analog Scale, from 0 to 100 mm, where 0 = no pain and 100 = worst imaginable pain
Time Frame: 12 months
Population: Intention-to-Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Evoke SCS With Feedback | Evoke SCS With Conventional
Number analyzed (Participants) | 59 | 59
Participants | 47 | 34
Statistical Analysis 1: Comparison: Evoke SCS With Feedback vs Evoke SCS With Conventional; Test type: Non-Inferiority — non-inferiority margin (δ) of 10%; p < 0.001, normal approximation to the binomial — significance threshold (α) of 0.05

ADVERSE EVENTS:
Time Frame: Through primary completion (3-months post-implant).
Description: Serious adverse event is an AE that
  * Led to death
  * Led to serious deterioration in the health of the subject and either resulted in a:
    1. life-threatening illness or injury or
    2. permanent impairment of a body structure or a body function or
    3. prolonged hospitalization or
    4. medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or a body function
  * Led to fetal distress, fetal death or congenital anomaly or birth defect
Arm/Group | Evoke SCS With Feedback | Evoke SCS With Conventional
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/67
Serious Adverse Events (participants affected / at risk) | 7/67 | 4/67
Other Adverse Events (participants affected / at risk) | 14/67 | 15/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Evoke SCS With Feedback (N=67) | Evoke SCS With Conventional (N=67)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Arrhythmia and Irregularities (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Chest Pain (Cardiac disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diverticulitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Epidural Abscess (Infections and infestations) | 0 (0) | 1 (1)
Facet Cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lead Breakage/Fracture (Product Issues) | 0 (0) | 1 (1)
Liver Abscess (Hepatobiliary disorders) | 1 (1) | 0 (0)
Renal Insufficiency (Renal and urinary disorders) | 0 (0) | 1 (1)
Suicidal Ideation or Attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Transient Ischemic Attack (Vascular disorders) | 1 (1) | 0 (0)
Wound Infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Evoke SCS With Feedback (N=67) | Evoke SCS With Conventional (N=67)
Upper Respiratory Symptoms or Upper Respiratory Tract Infection (Infections and infestations) | 7 (9) | 5 (5)
Fall or Trip or Slip or Twist (Injury, poisoning and procedural complications) | 3 (3) | 6 (7)
Lead Migration (Product Issues) | 4 (4) | 3 (3)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI may not publish their site results until study completion and multicenter results are published, unless multicenter results are not submitted for publication within 12 months of study completion or they receive Sponsor authorization. PI must notify sponsor within 30 days of submitting their site results. Sponsor may require a delay of up to 90 days if determined patent applications need to be filed or confidential information removed.

DOCUMENTS (2):
  • Study Protocol (2018-08-06): https://cdn.clinicaltrials.gov/large-docs/29/NCT02924129/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-01): https://cdn.clinicaltrials.gov/large-docs/29/NCT02924129/SAP_001.pdf